CLINICAL TRIAL: NCT00935129
Title: Treatment Satisfaction of Using OmniPod System Compared With Conventional Insulin Pump in Adults With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: rmc005431ctil
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2011-02

CONDITIONS: Type 1 Diabetes
Keywords: Treatment satisfaction; OmniPod; Insulin pump; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OmniPod system (Experimental): At this arm patients will be treated with the OmniPod system for 12 weeks
  Interventions: Device: OmniPod system
- patient's conventional pump (Active Comparator): At this arm patients will be treated with their conventional pump for 12 weeks
  Interventions: Device: Patient's conventional pump

INTERVENTIONS:
Device: OmniPod system — Patients will be treated with the OmniPod system for 12 weeks
  Arms: OmniPod system
Device: Patient's conventional pump — patients will be treated with their conventional pump for 12 weeks
  Arms: patient's conventional pump

SUMMARY:
Randomized, two arms, open study in order to evaluate treatment satisfaction of using OmniPod system compared with conventional insulin pump in adults with type 1 diabetes.

The study will include two consecutive 12 weeks treatment periods. According to randomization, each patient will be treated consecutively with both treatment arms: 12 weeks with OmniPod system and than 12 weeks with patient's previous insulin pump or vice versa.

DETAILED DESCRIPTION:
A Randomized, two arms, open, crossover study in order to evaluate treatment satisfaction of using OmniPod system compared with conventional insulin pump in adults with type 1 diabetes.

The study will include two consecutive 12 weeks treatment periods. According to randomization, each patient will be treated consecutively with both treatment arms: 12 weeks with OmniPod system and than 12 weeks with patient's previous insulin pump or vice versa.

Study will consist of 4 clinic visits taking place at -2,0,12 and 24 weeks and additional 4 telephone visits taking place at 4,8,16 and 20 weeks. In addition, patients will be invited one week prior to visit 5 and visit 8 in order to insert a continuous glucose sensor. Patients will complete DTSQ and Comfort & Function questionnaires at weeks 0, 12 and 24, before and at the end of each study arm.

On each clinical visits the following parameters will be evaluated: vital signs, HbA1c, 4 and 7 points glucose profile, hypoglycemia events, hyperglycemia events and pump related technical problems.

The telephone visits will include pump related technical problems solving and AE/SAE reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes diagnosed at least 1 year prior to study entry
2. Use of continuous subcutaneous insulin infusion therapy for at least one year
3. Age: 18-35 years old
4. HbA1c >8.0
5. At least 4 self blood glucose measurements per day
6. No more than one severe hypoglycaemic or ketoacidosis episode within the past year and none within the past month
7. Capable of reading pump screen in English
8. Able to understand and sign subject informed consent forms

Exclusion Criteria:

1. Any significant disease or conditions, including psychiatric disorders that in the opinion of the principal investigator are likely to effect subject compliance or the subjects ability to complete the study.
2. Patients participating in other device or drug studies
3. Clinical diagnosis of hypoglycaemic unawareness
4. Known dermal hypersensitivity to products that contain medical adhesive
5. Taking prescription medications that could complicate the management of glycemic control.
6. Inability to understand/complete the Treatment satisfaction questionnaire

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Treatment satisfaction | Diabetes Treatment Satisfaction Questionnare (DTSQ) will be completed at baseline, 12 and 24 weeks

SECONDARY OUTCOMES:
Comfort and function | Comfort and function questionnaires will be completed at weeks 0,12 and 24.
HbA1C | HbA1C will be measured at screening, baseline, 12 weeks and 24 weeks
Fructosamine | Fructosamine will be measured at baseline,12 and 24 weeks
7 points glucose profile | diary will be completed before every clinical visit
Pump related technical difficulties | pump related technical difficulties will be analyzed every telephone visit
continuous glucose measurements | continuous glucose sensor will be inserted one week before visits 5 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Principal Investigator — Rabin Medical Center
Locations (1):
- Schnider children's medical center, Petah Tikva, Israel

REFERENCES:
- [Derived] Lebenthal Y, Lazar L, Benzaquen H, Shalitin S, Phillip M. Patient perceptions of using the OmniPod system compared with conventional insulin pumps in young adults with type 1 diabetes. Diabetes Technol Ther. 2012 May;14(5):411-7. doi: 10.1089/dia.2011.0228. Epub 2012 Jan 27. PMID 22283640